CLINICAL TRIAL: NCT06669637
Title: Amplify EP Registry
Acronym: AMP
Status: Not yet recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: Amplify
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; Radiofrequency
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing AF Ablation using TactiFlex catheter: patients undergoing de novo or redo AF ablation procedures using TactiFlex ablation catheter following patients up to 6 to 12 months follow up.
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Ablation procedure for Atrial Fibrillation

SUMMARY:
An observational, prospective, multi-center, non-randomized registry designed to obtain real world clinical experience with the TactiFlex Catheter Ablation system in the treatment of Atrial Fibrillation. Patient assessments will occur at pre procedure and procedure, and 1 year post ablation

ELIGIBILITY:
Inclusion Criteria:

* Patients who, in the opinion of the investigator, are candidates for ablation to treat atrial fibrillation.
* Plans to undergo an ablation procedure using the TactiFlex Ablation Catheter™, Sensor Enabled™ (TactiFlex SE) manufactured by Abbott.
* De Novo or redo AF catheter ablation procedures.
* Able and willing to participate in baseline and all follow up evaluations.
* 18 years of age or older.

Exclusion Criteria:

* Enrolled in any other cardiac device clinical trial, investigational drug trial, or any other trial that may confound the results of the ablation procedure.
* In the opinion of the investigator, any known contraindication to an ablation procedure or to any device or drug required for use during an ablation procedure as assessed by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with atrial fibrillation undergoing ablation at selected sites who meet eligibility. Site in US, Canda, and OUS
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-11-22 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Long term effectiveness | 12-month
  defined as freedom from recurrence of AF/AT/AFL >30 sec at 12-month follow-up

SECONDARY OUTCOMES:
Acute success | at time of procedure
  ability to obtain pulmonary vein isolation during the ablation using TactiFlex catheter only
Acute safety | 30 days
  rate of acute safety events defined as procedure or device related complications that occur within 7 days of the procedure and incidence per-procedural complications that occur greater than 7 days but less than 30 days post ablation
Long term safety | 12 months
  Rate of long-term safety events defined as procedure or device related complications that occur greater than 30 days post ablation.

IPD SHARING:
Plan to Share IPD: No